CLINICAL TRIAL: NCT03461198
Title: A Single Center, Prospective, Open-label, Clinical Trial Using Micro-injections of Transparent Hyaluronic Acid Gel (Restylane® Silk) for Rejuvenation of the Aging Cheek
Brief Title: Micro-injections of Transparent Hyaluronic Acid Gel (Restylane® Silk) for Rejuvenation of the Aging Cheek
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Goldman, Butterwick, Fitzpatrick and Groff (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Restylane Silk Microinjections
Record Dates: First submitted 2018-03-05; First posted 2018-03-09 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Wrinkle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Treatment (Experimental): Restylane® Silk to a defined area of mid to low cheeks.
  Interventions: Device: Restylane® Silk

INTERVENTIONS:
Device: Restylane® Silk — Restylane® Silk to a defined area of mid to low cheeks

SUMMARY:
The objective of this study is to determine the efficacy and safety of Restylane® Silk microinjections when used in a grid-like injection pattern for the correction of fine lines to the cheeks.

DETAILED DESCRIPTION:
This is a single center, prospective, open-label, clinical trial using micro-injections of Restylane® Silk for correction of mid to low cheek fine lines and wrinkles. Twenty (20) subjects will be enrolled. Each subject will receive Restylane® Silk to a defined area of mid to low cheeks. The injections will be delivered intradermally via multiple 0.02 cc microinjections distributed in a grid array pattern with 1 cm between each injection point. A total surface area of 9-15 cm2 per cheek will be treated depending on the extent of fine lines in each subject. Following completion of injection treatment, manual massage will be applied to the full area to promote even distribution of the product. Each subject will undergo a total of three treatment sessions, one month apart, day 1, week 4, and week 8. The maximum amount of Restylane to be used per treatments session/per cheek is 1.5cc (not to exceed a total of 9 cc) per treated patient. Three dimensional digital photography utilizing the Vectra 3D System (Canfield) will be utilized to document pre-treatment status, sites of injection, and post-treatment effect. Subjects will be followed up at 4 weeks, 8 weeks, post-treatment day 90, and day 180.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female in general good health age 18 or over.
2. Mild to moderate static rhytids involving at least a 9 cm2 area of the mid to low cheeks.
3. Must be willing to give and sign a HIPPA form, photo consent and informed consent form.
4. Must be willing to comply with study dosing and complete the entire course of the study.
5. Female patients will be either of non-childbearing potential defined as:

   1. Having no uterus
   2. No menses for at least 12 months. Or;

   (WOCBP) women of childbearing potential must agree to use an effective method of birth control during the course of the study, such as:
   1. Oral contraceptive pill, injection, implant, patch, vaginal ring, intrauterine device
   2. Intrauterine coil
   3. Bilateral tubal ligation
   4. Barrier method used with an additional form of contraception (e.g., sponge, spermicide or condom)
   5. Abstinence (If practicing abstinence must agree to use barrier method described above (4) if becomes sexually active).
   6. Vasectomized partner (must agree to use barrier method described above (4) if becomes sexually active with un-vasectomized).
6. Negative urine pregnancy test results Baseline prior to study entry (if applicable)

Exclusion Criteria:

1. Pregnant, planning pregnancy during the course of the study or breastfeeding
2. Severe static rhytids to the mid to low cheeks
3. Previous use of any form of soft tissue augmentation in the treatment area within the past 12 months
4. Pre-existing medical or dermatologic condition in the treatment area that may affect the treatment or interpretation of treatment effect (at investigator discretion)
5. Presence of tattoo and/or scar in the treatment area that in the investigators opinion would interfere with study assessments
6. Use of oral/topical retinoids within 1 month of Baseline
7. Previous use of botulinum toxins in the treatment area within the past 6 months
8. Previous surgical procedure in the treatment area within the past 12 months
9. Presence or evidence of any conditions that in the opinion of the investigator might impede the subject's ability to give consent or comply with protocol requirements.
10. Current participation or participation within 30 days prior to the start of this study in a drug or other investigational research study
11. History of non-compliance with clinical research protocols
12. Ablative laser resurfacing to on their face within 12 months
13. Non-ablative laser or light procedures to their face within the past 3 months
14. Known allergy to Restylane® Silk or any of its constituents

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-02-26 (Actual); Primary Completion 2020-04-01 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy | Baseline to Day 180 post treatment
  Improvement on a validated 9-point Goldman-Fitzpatrick Wrinkle Scale (GFWS)

CONTACTS AND LOCATIONS:
Overall Officials: Mitchel P Goldman, MD, Principal Investigator — Cosmetic Laser Dermatology
Locations (1):
- Cosmetic Laser Dermatology, San Diego, California, United States